CLINICAL TRIAL: NCT04278274
Title: A Post-Neoadjuvant Treatment MRI Based AI System to Predict Pathologic Complete Response for Patients With Rectal Cancer: A Multicenter, Prospective Clinical Study
Brief Title: Post-Neoadjuvant Treatment MRI Based AI System to Predict pCR for Rectal Cancer
Acronym: MR-AI-pCR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); The Third Affiliated Hospital of Kunming Medical College. (Other)
Responsible Party: Principal Investigator, wanxiangbo, professor of Radiation Oncology, Vice Director, Department of Radiation Oncology, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: MR-AI-pCR 2020
Record Dates: First submitted 2020-02-19; First posted 2020-02-20 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Rectal Cancer
Keywords: Radiomics features; Artificial intelligence model; Locally advanced rectal cancer; Pathologic complete response; Neoadjuvant treatment
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients will be evaluated by artificial intelligence system and expert radiologist: the patients with locally advanced rectal cancer (LARC) finished the neoadjuvant treatment, and not yet receive total mesorectum excision (TME) surgery will be enrolled. The post-neoadjuvant treatment MRI images features of each enrolled patients will be captured by the artificial intelligence system, and evaluated by experienced radiologists as well. Blind to the pathologic report of TME specimen, both approaches further respectively yield a predicted pathologic response to neoadjuvant treatment for each enrolled patient, shown as pCR or non-pCR.
  Interventions: Procedure: artificial intelligence prediction system; Procedure: the radiologists

INTERVENTIONS:
Procedure: artificial intelligence prediction system — The tumor ROI in the post- neoadjuvant treatment MRI images will be manually delineated, and further subjected to the AI prediction system arm to verify the predictive accuracy of this AI prediction system in identifying the pCR individuals from non-pCR patients with LARC.
Procedure: the radiologists — The enrolled patients will be assigned to the trained experienced radiologists to evaluate their predictive accuracy in identifying the pCR individuals from non-pCR patients

SUMMARY:
In this study, investigators seek for a better way to identify the potential pathologic complete response (pCR) patients form non-pCR patients with locally advanced rectal cancer (LARC), based on their post-neoadjuvant treatment Magnetic Resonance Imaging (MRI) data.

Previously, a post neoadjuvant treatment MRI based radiomics AI model had been constructed and trained. Here, the predictive power of this artificial intelligence system and expert radiologist to identify pCR patients from non-pCR LARC patients will be compared in this prospective, multicenter, back-to-back clinical study

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational clinical study for seeking out a better way to predict the pathologic complete response (pCR) in patients with locally advanced rectal cancer (LARC) based on the post-neoadjuvant treatment Magnetic Resonance Imaging (MRI) data. Patients who have been pathologically diagnosed as rectal adenocarcinoma and defined as clinical II-III stage will be enrolled from the Sixth Affiliated Hospital of Sun Yat-sen University, Sir Run Run Shaw Hospital and the Third Affiliated Hospital of Kunming Medical College. All participants should follow a standard treatment protocol, including neoadjuvant treatment, total mesorectum excision (TME) surgery. Patients with LARC who received neoadjuvant treatment will be enrolled and their post-neoadjuvant treatment MRI images will be used to predict their pathologic response (pCR vs. non-pCR). The artificial intelligence prediction system and the expert radiologist will define the pathologic response as pCR or non-pCR, respectively. The pathologist will provide the final pathology report of TME surgery specimen (pCR or non-pCR) as a standard. The predictive efficacy of these two back-to-back approaches generated will be compared in this multicenter, prospective clinical study.

ELIGIBILITY:
Inclusion Criteria:

* pathologically diagnosed as rectal adenocarcinoma
* defined as clinical II-III staging (≥T3, and/or positive nodal status) without distant metastasis
* receive neoadjuvant chemoradiotherapy or chemotherapy
* pre- and post-neoadjuvant treatment MRI data obtained
* receive total mesorectum excision (TME) surgery after neoadjuvant therapy and get the pathologic assessment of tumor response

Exclusion Criteria:

* with history of other cancer
* insufficient imaging quality of MRI to delineate tumor volume or obtain measurements (e.g., lack of sequence, motion artifacts)
* not completing neoadjuvant chemotherapy or chemoradiotherapy
* tumor recurrence or distant metastasis during neoadjuvant treatment
* not undergoing surgery resulting in lack of pathologic assessment of tumor response

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the study, the population are the patients with LARC, who receive neoadjuvant chemoradiotherapy or chemotherapy and TME surgery. The response of neoadjuvant treatment is unknown.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2020-02-08 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
The area under curve (AUC) of Receiver Operating Characteristic (ROC) curves of AI prediction system and expert radiologists in prediction tumor response | baseline
  The area under curve (AUC) of Receiver Operating Characteristic (ROC) curves of AI prediction system and expert radiologists in identifying the pCR candidates from non-pCR individuals among neoadjuvant chemotherapy or chemoradiotherapy treated LARC patients will be calculated respectively.

SECONDARY OUTCOMES:
The specificity of AI prediction system and expert radiologists in prediction tumor response | baseline
  The specificity of AI prediction system and expert radiologists in identifying the pCR candidates from non-pCR individuals among neoadjuvant chemotherapy or chemoradiotherapy treated LARC patients will be calculated respectively.
The sensitivity of AI prediction system and expert radiologists in prediction tumor response | baseline
  The sensitivity of AI prediction system and expert radiologists in identifying the pCR candidates from non-pCR individuals among neoadjuvant chemotherapy or chemoradiotherapy treated LARC patients will be calculated respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbo Wan, MD, PhD, Study Chair — Sixth Affiliated Hospital, Sun Yat-sen University; Weidong Han, MD, PhD, Principal Investigator — Sir Run Run Shaw Hospital; Zhenhui Li, MD, Principal Investigator — The Third Affiliated Hospital of Kunming Medical College.
Locations (3):
- China (3):
  - the Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Kunming Medical College, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No